CLINICAL TRIAL: NCT01953484
Title: Changes in Spontaneous Ventilation in Response to Changes in Extracorporeal Carbon Dioxide Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VECLA-ECMO
Record Dates: First submitted 2013-09-09; First posted 2013-10-01 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

ARMS (3):
- Acute Respiratory Distress Syndrome (Experimental): Acute hypoxemia, bilateral pulmonary infiltrates and no evidence of primary left atrial hypertension
  Interventions: Other: Change in extracorporeal carbon dioxide removal
- Chronic Obstructive Pulmonary Disease (Experimental): Acute-on-Chronic Respiratory Insufficiency (patients with Chronic Obstructive Pulmonary Disease)
  Interventions: Other: Change in extracorporeal carbon dioxide removal
- Bridge to Lung Transplant (Experimental): Acute-on-Chronic Respiratory Insufficiency (patients awaiting lung transplant)
  Interventions: Other: Change in extracorporeal carbon dioxide removal

INTERVENTIONS:
Other: Change in extracorporeal carbon dioxide removal

SUMMARY:
In physiological conditions, spontaneous ventilation is controlled by blood carbon dioxide (and pH) levels. In healthy animals, extracorporeal carbon dioxide removal leads to hypoventilation or apnea (Kolobow et al., 1977). During acute respiratory insufficiency, extracorporeal carbon dioxide removal may be used to control spontaneous ventilation, limiting risks of lung damage and relieving dyspnea (Crotti et al., 2012). However, little is known about how spontaneous ventilation changes in response to changes in extracorporeal carbon dioxide removal during acute respiratory insufficiency, especially in humans.

Aim of this study is to monitor changes in spontaneous ventilation in awake patients treated with extracorporeal gas exchange support because of acute respiratory insufficiency, in response to changes in extracorporeal carbon dioxide removal.

ELIGIBILITY:
Inclusion Criteria:

* Acute Respiratory Insufficiency
* Extracorporeal gas exchange support
* The patient is spontaneously breathing (including assisted ventilation)

Exclusion Criteria:

- age below 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Spontaneous ventilation | 30-60 minutes after changing extracorporeal carbon dioxide removal
  Extracorporeal carbon dioxide removal will be increased or decreased changing the gas flow to the extracorporeal membrane lung. Actual extracorporeal carbon dioxide removal will be measured. Spontaneous respiratory rate, tidal volume, minute ventilation, esophageal pressure swings and comfort of the patient will be recorded 30-60 minutes after changing extracorporeal carbon dioxide removal.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan, Italy